CLINICAL TRIAL: NCT05731453
Title: Clinical Pilot Study for Personalized Risk-based Breast Cancer Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 494936
Record Dates: First submitted 2023-01-10; First posted 2023-02-16 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: risk based screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polygenetic risk score (Experimental): Assessment of polygenetic risk score for breast cancer
  Interventions: Genetic: Polygenetic risk score

INTERVENTIONS:
Genetic: Polygenetic risk score — Polygenetic risk score assessment for breast cancer

SUMMARY:
The study aims to evaluate the impact of implementing population-based genetics testing strategy for breast cancer precision prevention using the polygenic risk score and monogenic pathogenic variant (MPV) testing in the Norwegian healthcare setting.

DETAILED DESCRIPTION:
The study will recruit women age 40-50 referred for clinical mammography at the Vestre Viken Breast Center, with mammographic density BI-RADS a or d. After informed consent, saliva from the participants will be sampled and tested for polygenetic risk score (PRS) for breast cancer. The participants will be recommended future mammographic screening based on the PRS (standard screening, or more frequent/start at earlier age). The participants family history of cancer will be assessed, and if indicated, the participants will be referred for full genetic counselling/testing. The study will follow the women for 10 years for development of breast cancer as well as compliance to the recommended follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Women referred for clinical mammography in the Vestre Viken Breast Centre
* Breast density BI-RADS a or d
* 40-50 y.o.

Exclusion Criteria:

* Prior history of breast cancer or premalignant breast disease
* Prior genetic counselling/testing

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2035-11-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of breast cancer risk by polygenetic risk score in the study population | 10 years
  Polygenetic breast cancer risk score (PRS) as a numeric value with 10 percentile, as absolute 10-year breast cancer risk, and as relative risk compared with average women at the same age

SECONDARY OUTCOMES:
Compliance to individual recommedations for breast cancer screening | 10 years
  Percentage and frequencies of participants following their individual screening recommendations
Correlation of polygenetic risk score and breast cancer risk assessed by family history | 10 years
  Distribution of PRS among participants with increased breast cancer risk based on family history
Participants´ experience with study participation | 10 years
  Questionnaries on experience with the sampling process and feedback on a categorical scale (totally disagree, disagree, neutral, agree, totally agree)

CONTACTS AND LOCATIONS:
Overall Officials: Tone Hovda, Phd, Principal Investigator — Vestre Viken HT
Locations (1):
- Vestre Viken Hospital Trust, Drammen, Norway

IPD SHARING:
Plan to Share IPD: No